CLINICAL TRIAL: NCT06120504
Title: An Open-label Phase 1 Study to Evaluate the Safety of PF-08046045/SGN-35T in Adults With Advanced Malignancies
Brief Title: A Safety Study of PF-08046045/SGN-35T in Adults With Advanced Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated as part of strategic considerations
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGN35T-001; C5811001 (Other: Alias Study Number); 2022-502390-41-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Hodgkin Disease; Lymphoma, T-Cell, Peripheral; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin
Keywords: cHL; ALCL; PCL; PTCL; DLBCL; CTCL; Non-Hodgkin Lymphoma; Seattle Genetics
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Hodgkin Disease; Lymphoma, T-Cell, Peripheral; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-08046045 (Experimental): monotherapy
  Interventions: Drug: PF-08046045

INTERVENTIONS:
Drug: PF-08046045 — Given into the vein (IV; intravenously)
  Other Names: SGN-35T

SUMMARY:
This clinical trial is studying lymphoma. Lymphoma is a cancer that starts in the blood cells that fight infections. There are several types of lymphoma. This study will enroll people who have lymphoma, such as classical Hodgkin lymphoma, peripheral T-cell lymphoma including systemic anaplastic large cell lymphoma, diffuse large B-cell lymphoma, or some types of primary cutaneous lymphoma.

This clinical trial uses a drug called PF-08046045/SGN-35T. The study drug is in testing and has not been approved for sale. This is the first time PF-08046045 will be used in people. The study drug will be given as an infusion through a vein.

This study will test the safety of PF-08046045 in participants with lymphoma. It will also study the side effects of this drug. A side effect is anything a drug does to the body besides treating the disease.

This study will have three parts. Parts A and B of the study will find out the best dose and dosing schedule for PF-08046045. Part C will use the dose found in parts A and B to find out how safe PF-08046045 is and if it works to treat select lymphomas.

DETAILED DESCRIPTION:
This is a phase 1, open-label, multicenter study designed to characterize the safety, tolerability, pharmacokinetics, pharmacodynamics, and antitumor activity of PF-08046045/SGN-35T in adults with select relapsed/refractory lymphomas. PF-08046045 is a CD30-directed antibody-drug conjugate and will be studied in patients with lymphomas expressing CD30.

ELIGIBILITY:
Inclusion Criteria:

* Disease indication

  * For dose escalation and dose optimization (Part A and Part B):

    * Participants with a histologically confirmed lymphoid neoplasm (including relapsed/refractory [R/R] classical Hodgkin lymphoma [cHL], R/R peripheral T-cell lymphoma [PTCL], R/R systemic anaplastic large cell lymphoma [sALCL] , R/R mature B-cell neoplasms, and select R/R primary cutaneous lymphomas [PCLs]) who in the judgment of the investigator have no appropriate standard therapy available at the time of enrollment and are a candidate for PF-08046045 treatment.
    * Participants must have a detectable CD30 expression level (≥1%) in tumor tissue (except cHL and ALCL where CD30 is universally expressed).
  * For dose expansion (Part C)

    * Participants are eligible irrespective of CD30 expression on tumor tissue.
    * Participants with cHL: Participants with R/R cHL who have received at least 3 prior systemic therapies (autologous stem cell transplant [ASCT] and the associated high dose chemotherapy prior to ASCT are considered to be 1 prior line, along with post-transplant consolidation if progression has not occurred between transplant and start of consolidation) and meet all of the following additional criteria:

      * Participants who have not received ASCT must have refused or been deemed ineligible.
      * Participants must have received or been ineligible to receive an anti-PD-1 agent.
    * Participants with PTCL:

      * Participants with R/R PTCL (excluding R/R sALCL) who have received at least 2 prior systemic therapies or received at least 1 prior systemic therapy and there is no other available treatment that is considered appropriate by the investigator.
      * Participants with R/R sALCL must have ALK status documented and must meet one of the following criteria:

        * Disease recurrence or progression following at least 2 prior systemic therapies where 1 regimen included brentuximab vedotin, or
        * Disease recurrence or progression following only 1 prior line of therapy which included brentuximab vedotin, cyclophosphamide, doxorubicin, and prednisone
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score ≤1.
* Fluorodeoxyglucose positron emission tomography (FDG PET) avid and bidimensional measurable disease as documented by radiographic technique (spiral CT preferred) per Lugano criteria at baseline (Cheson 2014) (not applicable for subjects with PCL).

Exclusion Criteria:

* Participants who have received more than 2 prior brentuximab vedotin-based lines of therapy.
* History of another malignancy within 3 years before the first dose of study intervention, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death.
* Active cerebral/meningeal disease related to the underlying malignancy.
* Received previous ASCT infusion <12 weeks prior to first PF-08046045 dose.
* Participants with previous allogeneic stem cell transplant (SCT) if they meet any of the following criteria:

  * <100 days from allogeneic SCT. Participants ≥100 days from allogeneic SCT who are stable without immunosuppressive therapy for at least 12 weeks are permitted.
  * Active acute or chronic graft versus host disease or receiving immunosuppressive therapy as treatment for or prophylaxis against graft versus host disease.
* Participants with previous allogeneic SCT and participants considered at high risk for CMV reactivation (eg, recent prior CAR-T or bispecific antibody therapy) if they meet the following criteria: Cytomegalovirus (CMV) PCR ≥500 IU/mL, OR rising DNA levels >5-times baseline within 1 month, OR detectable CMV PCR receiving pre-emptive therapy; prior PCR positivity that was successfully treated is acceptable provided the baseline PCR result is negative prior to the first dose of study intervention.
* Grade 2 or higher pulmonary disease unrelated to underlying malignancy, or history of Grade 2 or higher drug-induced interstitial lung disease (ILD) or immune checkpoint inhibitor (ICI)-related ILD.
* Clinically significant lung disease requiring systemic corticosteroid treatment within 6 months prior to enrollment or who are suspected to have such diseases via radiographic imaging and/or functional tests conducted during the screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30-37 days after last study treatment, approximately 1 year
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention
Number of participants with laboratory abnormalities | Through 30-37 days after last study treatment, approximately 1 year
Number of participants with dose modifications due to AEs | Up to approximately 1 year
Number of participants with dose-limiting toxicities (DLTs) | Up to 21 days
Number of participants with DLTs by dose level | Up to 21 days

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter - Area under the concentration-time curve (AUC) | Through 30-37 days after last study treatment, approximately 1 year
  To be summarized using descriptive statistics
PK parameter - Maximum concentration (Cmax) | Through 30-37 days after last study treatment, approximately 1 year
  To be summarized using descriptive statistics
PK parameter - Time to Cmax (Tmax) | Through 30-37 days after last study treatment, approximately 1 year
  To be summarized using descriptive statistics
Number of participants with antidrug antibodies (ADA) | Through 30-37 days after last study treatment, approximately 1 year
  To be summarized using descriptive statistics
Objective response rate (ORR) as assessed by the investigator | Up to approximately 1 year
  A subject is determined to have an objective response if, based on disease-specific assessment criteria, they achieve a complete response (CR) or partial response (PR) as assessed by the investigator. The ORR is defined as the percentage of participants with an objective response.
Complete response (CR) rate as assessed by the investigator | Up to approximately 1 year
  CR rate is defined as the percentage of subjects with CR.
Duration of response (DOR) | Up to approximately 1 year
  DOR is defined as the time from the start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression per disease-specific assessment criteria as assessed by the investigator or to death due to any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (16):
  - Stanford Cancer Center / Blood and Marrow Transplant Program, Palo Alto, California
  - University of Miami Hospital and Clinics - Lennar, Coral Gables, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - University of Miami, Miami, Florida
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - MSK Monmouth., Middletown, New Jersey
  - MSK Bergen., Montvale, New Jersey
  - Hackensack University Medical Center (From Road), Paramus, New Jersey
  - MSK Commack., Commack, New York
  - MSK Westchester., Harrison, New York
  - Memorial Sloan Kettering Cancer Center-Investigational Drug Service Pharmacy, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - Memorial Sloan Kettering Cancer Center-Main Campus, New York, New York
  - MSK Nassau., Uniondale, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Hospital Universitario Fundacion Jimenez Diaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGN35T-001